CLINICAL TRIAL: NCT02323906
Title: A Phase 1b, Multi-Center, Open-Label, Dose Finding Study of CC-122 in Combination With Sorafenib in Subjects With Unresectable Hepatocellular Carcinoma
Brief Title: Safety and Efficacy Study of CC-122 Combined With Sorafenib for Primary Liver Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment and business decision. No safety concerns were identified for the study drugs.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-122-HCC-001
Record Dates: First submitted 2014-11-24; First posted 2014-12-24 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular; Carcinoma; Phase 1; CC-122; Sorafenib,; Nexavar; Unresectable Hepatocellular Carcinoma; Unresectable HCCAdvanced,; Hepatocellular Carcinoma; liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma; Liver Neoplasms | interventions — 3-(5-amino-2-methyl-4-oxoquinazolin-3(4H)-yl)piperidine-2,6-dione; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CC-122 + Fixed-dose Sorafenib (Experimental): A dose escalation and expansion clinical study of CC-122 in combination with sorafenib in subjects with unresectable HCC who have received no prior systemic therapy for HCC.
  The dose escalation part of the study will explore several dose levels of CC-122 in combination with sorafenib, followed by an expansion part.
  Interventions: Drug: CC-122; Drug: Sorafenib

INTERVENTIONS:
Drug: CC-122 — Investigational new drug
Drug: Sorafenib — Kinase inhibitor
  Other Names: Nexavar

SUMMARY:
CC-122-HCC-001 is a Phase 1b dose escalation and expansion clinical study of CC-122 in combination with sorafenib for subjects with unresectable HCC who have received no prior systemic therapy for HCC. The dose escalation phase of the study will explore several dose levels of CC-122 in combination with sorafenib, followed by an expansion part of the study using the optimal combination dose regimen.

DETAILED DESCRIPTION:
The primary objective of the study is to determine the safety and tolerability of CC-122 administered orally in combination with sorafenib, and to define the non-tolerated dose (NTD), the maximum tolerated dose (MTD), and the recommended phase 2 dose (RP2D).

The secondary objective of the study is to determine the preliminary efficacy of CC-122 in combination with sorafenib, based on response Evaluation Criteria in Solid Tumors (RECIST 1.1)

ELIGIBILITY:
Inclusion Criteria:

1. Subject understands and voluntarily signs an informed consent document prior to conducting any study related assessments/procedures
2. Subject is 18 years of age or more at the time of signing the Informed Consent Form
3. Subject has a confirmed pathologic diagnosis of Hepatocellular carcinoma according to the American Association for the Study of Liver Diseases Guidelines.A biopsy performed at screening may serve as a diagnostic biopsy for subjects with radiographic diagnosis.
4. Subject has unresectable stage B (intermediate), or C (advanced) Hepatocellular carcinoma according to the Barcelona Clinic Liver Cancer staging.Stage B subjects must have progressed after, or are not eligible for curative resection, transplantation, embolic, or ablative therapies
5. Subject has at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors version 1.1. Evaluable target lesions may not have been treated with local therapy; previously treated lesions may only be evaluated as target lesions if they are the only lesions available and have shown objective definite progression after prior treatment. Local therapy must have been completed at least four weeks prior to baseline tumor evaluation
6. Satisfactory archival tumor biopsy tissue is retrieved, or new tumor biopsy is performed, prior to starting Cycle 1
7. Subject has life expectancy of more than 12 weeks
8. Subject has Eastern Cooperative Oncology Group Performance Status of 0 or 1
9. Subject has Child-Pugh score of less than 7 (ie, class A or better) with neither encephalopathy nor clinically significant ascites (ascites requiring paracentesis within 3 months of signing the ICF is excluded). Child-Pugh status is calculated based on clinical findings and laboratory results during the screening period.
10. Subject has the following laboratory parameters at screening:

    Adequate hematologic function including:
    1. Absolute Neutrophil Count of at least 1.5 x 109/L
    2. Platelets of at least 75,000 x 106/L
    3. Hemoglobin of at least 9 g/dL
    4. International Normalized Ratio of at least 1.7

    Adequate hepatic function including:
    1. Serum aspartate aminotransferase and alanine amino-transferase of at least 5 times the upper limit of normal
    2. Serum total bilirubin of at least 3 mg/dL
    3. Serum albumin of at least 2.8 g/dL Note: Laboratories in combination must still be Child Pugh score less than 7

    Other laboratory parameters:
    1. Serum creatinine of at least 1.5 times the upper limit of normal
    2. Potassium within normal range or corrected with supplements
11. For subjects with known or suspected cirrhosis, esophagogastroduodenoscopy ) within 12 months of signing the informed consent form, showing no evidence of untreated varices or stigmata of active bleeding (such as active ulcer, visible vessel, or blood) is required.

    Subjects with history of upper GI bleeding must have an EGD of 3 months or less prior to signing the consent form confirming adequate prior endoscopic therapy (eg, no evidence of any untreated varices, recent or active bleeding, stigmata suggesting high risk for bleeding, active ulcer). Subjects with history/suspected esophageal varices must be on optimal medical management (eg, proton pump inhibitor and non-selective beta-blocker) per local institutional policy.
12. Subject is able to adhere to the study visit schedule and other protocol requirements
13. Pregnancy Prevention Risk Management Plan

    1. Females of childbearing potential must undergo pregnancy testing based on the frequency outlined in Pregnancy Prevention Risk Minimization Plan and pregnancy results must be negative.
    2. Unless practicing complete abstinence from heterosexual intercourse, sexually active FCBP must agree to use adequate contraceptive methods as specified in Pregnancy Prevention Risk Minimization Plan.

       * Complete abstinence is only acceptable in cases where this is the preferred and usual lifestyle of the subject.
       * Periodic abstinence (calendar ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable.
    3. Males (including those who have had a vasectomy) must use barrier contraception (condoms) when engaging in sexual activity with Female of Childbearing Potential as specified in Pregnancy Prevention Risk Minimization Plan.
    4. Males must agree not to donate semen or sperm for 3 months after last dose of CC-122.
    5. All subjects must:

       * Understand that CC-122 could have a potential teratogenic risk.
       * Agree to abstain from donating blood while taking CC-122 or sorafenib and following discontinuation of their use.
       * Agree not to share either study drug with another person.
    6. Other than the subject, Female of Childbearing Potential and males able to father a child should not handle CC-122 or touch the capsules, unless gloves are worn.
    7. Be counseled about pregnancy precautions and risks of fetal exposure

Exclusion Criteria:

* 1. Subject has received previous systemic therapy for Hepatocellular carcinoma including sorafenib, chemotherapy and investigational agents 2. Subject has received any local anticancer therapy ≤ 4 weeks prior to baseline tumor evaluation 3. Subject has undergone major surgery within the last 4 weeks or minor surgery within the last 2 weeks prior to signing the Informed Consent Form or who have not recovered from surgery 4. Subject has received an investigational drug or therapy for disease other than Hepatocellular carcinoma within the last 4 weeks or 5 half-lives, whichever is shorter, prior to signing the Informed Consent Form 5. Subject has completed any radiation treatment less than 2 weeks prior to signing the Informed Consent Form 6. Subject has received the last dose of α-interferon, ribavirin, sofobuvir and/or other antiviral therapies for Hepatitis C Virus (HCV) less than 4 weeks prior to signing the Informed Consent Form 7. Subject has any clinically significant bleeding, including bleeding from esophageal/gastric varices within ≤ 3 months of signing the informed consent form, which required transfusion, surgical procedure or hospitalization. Esophageal varices should be treated according to local standard practice (eg, ligation or banding and procedure completed ≤ 3 months prior to signing the informed consent form). See Inclusion Criterion 10 8. Subjects requiring therapeutic anticoagulation with either warfarin or low molecular weight heparin. Low dose low molecular weight heparin for catheter maintenance are permitted 9. Subject has tumor invasion of stomach or duodenum 10. Subject has histologic proof of fibrolamellar carcinoma 11. Subjects with known symptomatic brain metastasis 12. Subject has persistent diarrhea due to a malabsorptive syndrome (such as celiac sprue or inflammatory bowel disease) malabsorption ≥ National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE, Version 4.03) Grade 2, despite medical management, or any other significant GI disorder that could affect the absorption of either study drug 13. Subject has history of concurrent second cancers requiring active, ongoing systemic treatment. 14. Subject has a known history of human immunodeficiency virus (HIV) seropositivity (HIV testing is not mandatory) 15. Subject has peripheral neuropathy of at least NCI CTCAE Grade 2 16. Subject has a history of persistent skin rash of at least NCI CTCAE Grade 2 17. Subject has impaired cardiac function or clinically significant cardiac disease including any of the following:

  1. LVEF (left ventricular ejection fraction) of 45% or less as determined by MUGA (multi-gated acquisition) or ECHO (Echocardiogram)
  2. Complete left bundle branch or bifascicular block
  3. Congenital long QT syndrome
  4. Persistent or clinically meaningful ventricular arrhythmias
  5. QTcF greater than 460 msec on Screening ECG (mean of triplicate recordings)
  6. Unstable angina pectoris or myocardial infarction less than 6 months prior to starting either study drug
  7. Uncontrolled hypertension (blood pressure greater than 140/90 mmHg on at least 2 measurements on sequential visits, despite blood pressure medication)
* Subjects with baseline blood pressure 140/90 mmHg are eligible but must have optimal medication for blood pressure management h. Troponin-T value more than the upper limit of normal or BNP greater than 100 pg/mL 18. Subject has acute or chronic active infectious disorders or uncontrolled nonmalignant illnesses whose control, in the opinion of the investigator, may be jeopardized by complications of this study therapy. Chronic hepatitis B and C virus (HBV and HCV) are excepted (ie, eligible for study); HBV requires antiviral therapy 19. Subject has undergone liver transplantation or other solid organ transplantation requiring immunosuppression 20. Subject is receiving chronic treatment with systemic corticosteroids or other potentially immunosuppressive agent. Intermittent topical or local injection of corticosteroids and oral/IV aldosterone or other mineralocorticoids is allowed 21. Subjects with history of non-healing wounds or ulcers, or bone fractures less than 3 months of a prior fracture 22. Subject is being treated with concomitant strong CYP3A4 inducers such as St. John's Wort, dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, phenobarbital. The use of concomitant strong CYP3A4 inducers may decrease sorafenib plasma concentrations and must be avoided.

  23. Subject is a female who is pregnant or is breast feeding 24. Subject is unwilling or unable to comply with the protocol, in the opinion of the investigator 25. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study 26. Subject has any condition that confounds the ability to interpret data from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01-16 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Adverse Event | Up to 3 years
  Number of Participants with Adverse Events
Dose-Limiting Toxicity (DLT) | 28 Days
  Number of participants with a DLT. A DLT is defined as a treatment-related AE(s) occurring in Cycle 1 (including predose assessments on Cycle 2 Day 1).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 4 years
  Percentage of subjects with complete response or partial response using Response Evaluation Criteria in Solid Tumor (RECIST 1.1).
Disease control rate (DCR) | Up to 4 years
  Percentage of subjects with complete response, partial response or stable disease using Response Evaluation Criteria in Solid Tumor (RECIST 1.1).
Duration of response (DoR) | Up to 4 years
  Duration from the time of measurement criteria are first met for complete response or partial response until tumor progression using RECIST 1.1 or death.
Progression-free survival | Up to 4 years
  Number of participants who survive without tumor progression using RECIST 1.1and time from the first dose date until objective tumor progression or death, whichever occurs first.
Overall survival | Up to 4 years
  Number of participants who survive and the time from the first dose to death with any cause.
Time to progression (TTP) | Up to 4 years
  Number of participants who do not have tumor progression using RECIST 1.1 and the time from the first dose date until objective tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Hege, MD, Study Director — Celgene Corporation
Locations (8):
- United States (8):
  - University of California San Francisco, San Francisco, California
  - University of Florida College of Med, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Henry Ford Hospital, Detroit, Michigan
  - Greenville Hospital System, Greenville, South Carolina
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington